CLINICAL TRIAL: NCT03403660
Title: Physician Attire and Appreciation of Physician Communication in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB 17-0096
Record Dates: First submitted 2017-12-20; First posted 2018-01-18 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Patient Satisfaction
Keywords: Attire; White coat; Patient physician communication
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Women are randomly assigned to having their postpartum physician team wear a white coat (WC) or not (no-WC) during rounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non white coat rounding (Experimental): The postpartum physician rounding in this group will be performed wearing white coat.
  Interventions: Other: non White coat
- White coat rounding (Placebo Comparator): The postpartum physician rounding in this group will be performed not wearing white coat.
  Interventions: Other: non White coat

INTERVENTIONS:
Other: non White coat — Postpartum patients are randomized to either arm of the study (white coat or standard scrub suit only) by location. All the obstetric physicians associated with patient's postpartum care should use or not use white coat in every single encounter with patient.

SUMMARY:
Wearing white coat during hospital rounds has been associated with increased risk of colonization and transmission of resistant pathogens. On the other hand, studies have shown that physicians' attire affects patients' confidence in their physician and the patient-physician relationship. The results of these studies were highly dependent on the practice setting, with no data in postpartum patients.

The objective is to test the hypothesis that not wearing a white coat during physician postpartum rounds impact patient-physician communication scores.

DETAILED DESCRIPTION:
Patient satisfaction is an important measure of quality of care. One of the most important variables in patients satisfaction scores is the physician communication skills. There have been several studies evaluating different strategies to improve the patient perceptions of patient - physician communication including delayed physician rounds, improvement of handoff strategies, and family centered rounds. Additionally, research has shown that patients develop a first impression of their physician based on the physician's verbal and nonverbal communication, including the clothing and cleanliness. Patient - physician communication scores not only have an impact on patient care, but are also now linked to Medicare reimbursements.

White coats have been widely used in the medical profession, however some physicians believe that this can be a nonverbal barrier to patient's interaction. Prior studies on the impact of physician attire have reported conflicting results. In a survey published by Cha et al, obstetric and gynecologic patients seen in the outpatient clinic preferred that the resident use white coats. Another study showed that patients favor the use of white coat in the Internal Medicine outpatient clinic which may favorably influence trust and confidence in the medical encounter.

No randomized controlled trial has been published on the impact of the use of white coat on patient - physician communication scores in the postpartum patients. This trial's primary outcome is to evaluate the impact of physician attire (specifically wearing white coat) during postpartum rounds on "patient - physician communication" scores.

This study is a randomized controlled trial performed in postpartum patients to evaluate the impact of not wearing white coat during rounds on "patient - physician communication" scores.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18 years and <50 years
* Patient admitted to postpartum floor at University of Texas Medical Branch (UTMB)
* Patient care managed by obstetric physicians during the postpartum period.

Exclusion Criteria:

* Patient admitted to ICU
* Delivery resulting in stillbirth Patient not fluent in Spanish and/or English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Patient - physician communication score | 24 to 120 hours
  Obtained from the three Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) questions.

SECONDARY OUTCOMES:
Hospital rating scores | 24 to 120 hours
  Obtained from one question of the HCAHPS survey
Recommending the hospital to friends and family | 24 to 120 hours
  Obtained from one question of the HCAHPS survey
Physician attire rating score | 24 to 120 hours
  Rated from 1 to 4
White coat use | 24 to 120 hours
  Patient answer if she remember or not if their physician were using white coat.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio La Rosa, MD, Study Director — University of Texas
Locations (1):
- Universty of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No